CLINICAL TRIAL: NCT05046964
Title: Correlation of Non-invasive Hemoglobin Measurement With Bleeding During Cesarean Delivery: The PPHgb Study
Brief Title: The PPHgb Study: Non-Invasive Hemoglobin Measurement
Status: Completed | Type: Observational
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Jaclyn Phillips, Principal Investigator, George Washington University
Other Study IDs: NCR191913
Record Dates: First submitted 2021-06-23; First posted 2021-09-16 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Postpartum Hemorrhage
Keywords: hemoglobin
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Masimo Radical-7 Pulse CO-Oximeter — The Radical-7 Pulse CO-Oximeter uses photospectroscopy to non-invasively measure the total hemoglobin (SpHb) in a patient's blood throughout their C-section.

SUMMARY:
This project is a prospective observational study aimed to assess the use of non-invasive hemoglobin measurement in anticipating postpartum hemorrhage and predicting estimated blood loss. The non-invasive hemoglobin device is the Radical-7 Pulse CO-Oximeter which is a spectrophotometer manufactured by Masimo, Inc. Participants in the study will be undergoing a cesarean delivery at the George Washington University Hospital and during delivery the patient will wear the device on their fingertip so that hemoglobin measurements can be continuously recorded. No changes from routine medical management will occur during the study.

DETAILED DESCRIPTION:
This project is a prospective, observational study aimed to predict bleeding using hemoglobin trends measured non-invasively in patients undergoing elective cesarean delivery at the George Washington University Hospital.

The primary outcome is trend in hemoglobin measurement, at which additional interventions are required to control hemorrhage. The overall goal is to be able to determine a threshold point in which a drop in the hemoglobin level indicates severe bleeding in anticipation of postpartum hemorrhage. Through the observation of the continuous monitoring of hemoglobin across all participants and correlating those with severe hemorrhage to the magnitude of drop or time of drop, this could potentially optimize the hemorrhage protocol and might limit the need for blood transfusion and decrease maternal mortality and morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women age 18 - 50 years old
* Patients scheduled for cesarean delivery at >34 weeks gestation
* Patients who failed trial of labor and require cesarean delivery

Exclusion Criteria:

* Patients with spontaneous or operative vaginal delivery
* Patients with hemoglobinopathies (qualitative defects, sickle-cell anemia) and hemoglobin synthesis disorders (quantitative defects such as thalassemia)
* Patients with peripheral vascular diseases and skin conditions that affect blood vessels in the digit
* Patients with hyperbilirubinemia

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women between the age of 18 - 50 years old
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
Determine the critical threshold of SpHb drop during cesarean delivery | At the time of surgery
Correlation of the time a SpHb drop occurs with the time of hemorrhagic intervention decision | At the time of surgery
  Hemorrhagic interventions include: uterotonic drugs, surgical suturing, uterine tamponade devices, blood transfusion, etc.

SECONDARY OUTCOMES:
Correlation of the change in SpHb from pre-delivery to post-delivery values and the reported estimated blood loss or change in laboratory blood hemoglobin values. | Within 72 hours before surgery and 24 hours after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- The GW Medical Faculty Associates, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
Only aggregate de-identified information will be disclosed for this study